CLINICAL TRIAL: NCT00201734
Title: A Phase I Dose Escalation Study of Capecitabine, Carboplatin and Weekly Paclitaxel and a Phase II Trial of the Same Combination in Patients With Adenocarcinoma of Unknown Primary
Brief Title: Capecitabine, Carboplatin and Weekly Paclitaxel for Patients With Solid Tumors and Adenocarcinoma of Unknown Primary
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to lack of funding provided for Phase II portion of trial
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Tony Bekaii-Saab, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-0317; NCI-2011-03593 (Registry Identifier: Clinical Trials Reporting Program)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2016-06-01 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-08

CONDITIONS: Tumors; Unknown Primary Tumors; Adenocarcinoma
Keywords: Adenocarcinoma
MeSH Terms: conditions — Neoplasms; Neoplasms, Unknown Primary; Adenocarcinoma | interventions — Capecitabine; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive paclitaxel IV over 60 minutes on days 1, 8, and 15, carboplatin IV over 1-2 hours on day 1, and capecitabine PO BID on days 8-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Capecitabine; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Capecitabine — Level 1: 500 mg/m2 orally twice daily Days 8 - 21 of each cycle. Level 2: 750 mg/m2 orally twice daily Days 8 - 21 of each cycle. Level 3 - 5: 1000mg/m2 orally twice daily Days 8 - 21 of each cycle.
  Other Names: Xeloda
Drug: Carboplatin — Levels 1-5: AUC of 6 every 4 weeks.
  Other Names: Paraplatin; CBDCA
Drug: Paclitaxel — Level 1-3: 60 mg/m2/week. Level 4: 80 mg/m2/week. Level 5: 100 mg/m2/week.
  Other Names: Onxol; Taxol

SUMMARY:
This study will determine the maximum tolerated dose of the triplet combination of capecitabine that can be administered in combination with weekly paclitaxel and every four weeks with carboplatin.

DETAILED DESCRIPTION:
Rationale: The combination of the chemotherapy drugs paclitaxel and carboplatin is one of the most common combination regimens used in clinical practice for cancer. These agents are used for a variety of cancers. The current study builds on previous research about treatment schedules for administering these agents to reduce toxicity and optimize efficacy. The phase I and II portions of the current study combine paclitaxel and carboplatin with capecitabine in patients. Researchers are seeking to identify the highest dose of capecitabine and paclitaxel in combination with carboplatin for this patient population, as well as to gather information about preliminary efficacy.

Purpose: The phase I portion of this study will evaluate the maximum tolerated dose of capecitabine and paclitaxel in combination with carboplatin for patients. The phase II portion of this study will assess the objective response rate in patients using the same treatment combination. Toxicities will be closely measured in both phases of the study.

Treatment: Patients in this study will be given capecitabine, carboplatin, and paclitaxel. Capecitabine will be given through oral pills. Carboplatin and paclitaxel will be given through intravenous infusions. Treatment drugs will be given on a four-week cycle. Carboplatin will be administered on day 1, paclitaxel weekly for the first 3 weeks, and capecitabine twice daily on days 8 through 21 of each cycle. No treatments will be given during the fourth week of each treatment cycle. During the phase I portion of the study, patients may receive different doses of capecitabine and paclitaxel since the purpose is to identify the maximum tolerated dose of each drug in combination with carboplatin. Once the maximum tolerated dose of these agents is identified during phase I, the phase II portion of the study will begin. Treatments will be discontinued due to disease growth or unacceptable side effects. Several tests and exams will be given throughout the study to closely monitor patients.

ELIGIBILITY:
Inclusion Criteria for Phase I:

* All advanced solid malignancies
* Any prior chemotherapy permitted
* Performance Status 0-2

Inclusion Criteria for Phase II:

* Adenocarcinoma of unknown primary
* No prior chemo permitted
* Performance Status 0-2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2005-06; Primary Completion 2007-11 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tony Bekaii-Saab, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- [Background] Mikhail S, Lustberg MB, Ruppert AS, Mortazavi A, Monk P, Kleiber B, Villalona-Calero M, Bekaii-Saab T. Biomodulation of capecitabine by paclitaxel and carboplatin in advanced solid tumors and adenocarcinoma of unknown primary. Cancer Chemother Pharmacol. 2015 Nov;76(5):1005-12. doi: 10.1007/s00280-015-2877-6. Epub 2015 Sep 28. PMID 26416564
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled to the trial between July 2005 and November 2007
Groups:
- Phase I: Cycles will be of 4-week duration. Carboplatin was administered on day 1 intravenously for 3 weeks (days 1, 8, 15) and paclitaxel weekly intravenously for 3 weeks on days 1, 8 and 15. Capecitabine was given orally twice daily days 18-21 followed by 1 week rest.
- Phase II: Phase II trial combination at the recommended doses from the Phase I portion in patients with adenocarcinoma of unknown primary site.
Period: Overall Study
Arm/Group | Phase I | Phase II
Started | 32 | 25
Patients Not Evaluable | 3 | 0
Completed | 29 | 25
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I | Phase II | Total
Number analyzed (Participants) | 32 | 25 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 21 | 49
  >=65 years | 4 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 12 | 18
  Male | 26 | 13 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 29 | 24 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: patients]
  United States | 32 | 25 | 57

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose in Phase I Portion of Study
Description: Determine the maximum tolerated dose of the triplet combination of capecitabine that can be administered in combination with weekly paclitaxel and every four weeks carboplatin.
Time Frame: Every 3 weeks, for up to 24 weeks
Measure: Number; unit: mg/m2
Groups:
- Phase I Patients: Cycles will be of 4-week duration. Carboplatin was administered on day 1 intravenously for 3 weeks (days 1, 8, 15) and paclitaxel weekly intravenously for 3 weeks on days 1, 8 and 15. Capecitabine was given orally twice daily days 18-21 followed by 1 week rest.
Arm/Group | Phase I Patients
Number analyzed (Participants) | 29
mg/m2 | 750

2. Primary Outcome: Objective Response Rate (ORR) for the Phase II Portion of the Study. CR+PR Per RECIST v1.0 Criteria Using a Single Arm , Two Stage Minimax Design.
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Every 3 weeks, for up to 24 weeks
Population: The Phase II study was prematurely terminated at 25 patients due to cessation of funding
Measure: Number (95% Confidence Interval); unit: percent of patients
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 29 | 25
percent of patients | 21 [8 to 40] | 32 [15 to 54]

3. Secondary Outcome: Phase I: To Determine Side Effects
Description: The common clinically significant grade 3 and 4 toxicities graded using the National Cancer Institutes Common Toxicity Criteria version 3.0
Time Frame: Every 3 weeks, for up to 24 weeks
Population: Three patients enrolled on Phase I portion of trial were not evaluable for toxicity.
Measure: Number; unit: percent of patients
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 29 | 25
percent of patients
  Neutropenia | 86 | 72
  Thrombocytopenia | 72 | 72
  Fatigue | 76 | 84

4. Secondary Outcome: Progression-Free Survival at 6 Months for Patients
Description: For patients enrolled on the Phase II portion of the trial Progression Free Survival (PFS) was measured from the percentage of patients that were still alive, without evidence of disease progression for 6 months following the initiation of treatment. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: up to 6 years
Measure: Number (95% Confidence Interval); unit: percent of patients
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 0 | 25
percent of patients |  | 38 [22 to 54]

5. Secondary Outcome: One Year Survival for Patients
Description: For patients enrolled on the Phase II portion of the trial the One-year survival was measured as the percentage of patients alive 1 year after their treatment in the trial.
Time Frame: Up to 1 year
Measure: Number (95% Confidence Interval); unit: percent of patients
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 0 | 25
percent of patients |  | 44 [24 to 62]

6. Secondary Outcome: Time to Tumor Progression for Patients
Description: For patients enrolled on the Phase II portion of the trial the time to progression was measured as the time from when the patient started treatment to the time the patient is first recorded as having disease progression or the date of death if the patient dies due to causes other than disease progression.
Time Frame: Up to 6 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 0 | 25
months |  | 5.5 [2.8 to 10.8]

ADVERSE EVENTS:
Description: Adverse Events were graded using the National Cancer Institute Common Toxicity Criteria version 3.0.
Arm/Group | Phase I | Phase II
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/25
Other Adverse Events (participants affected / at risk) | 29/29 | 25/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (N=29) | Phase II (N=25)
Anemia (Blood and lymphatic system disorders) | 24 (24) | 22 (22)
Leukopenia (Blood and lymphatic system disorders) | 28 (28) | 10 (10)
Lymphopenia (Blood and lymphatic system disorders) | 19 (19) | 12 (12)
Neutropenia (Blood and lymphatic system disorders) | 25 (25) | 18 (18)
Thrombocytopenia (Blood and lymphatic system disorders) | 21 (21) | 18 (18)
Anorexia (Gastrointestinal disorders) | 10 (10) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 18 (18) | 18 (18)
Fatigue (General disorders) | 22 (22) | 21 (21)
Fever without Neutropenia (General disorders) | 8 (8) | 3 (3)
Hand Foot Syndrome (Skin and subcutaneous tissue disorders) | 13 (13) | 5 (5)
Mucositis (Gastrointestinal disorders) | 8 (8) | 11 (11)
Nausea (Gastrointestinal disorders) | 23 (23) | 18 (18)
Vomiting (Gastrointestinal disorders) | 11 (11) | 14 (14)
Neuropathy (Nervous system disorders) | 18 (18) | 15 (15)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes